CLINICAL TRIAL: NCT06368557
Title: Internet-based Cognitive Behavioral Intervention for Adolescents With Anxiety Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region of Southern Denmark (Other)
Collaborators: University of Aarhus (Other)
Responsible Party: Principal Investigator, Kim Mathiasen, Associate Professor, Region of Southern Denmark
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 22/59602
Record Dates: First submitted 2023-10-16; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Anxiety Disorders
Keywords: Adolescents; Anxiety Disorders; Cognitive behavioral therapy; Internet-based; Digital health
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The RCT is designed as a superiority RCT with the three conditions 1) iCBT with planned feedback 2) iCBT with on-demand feedback and 3) waitlist control. The allocation ratio is 1:1:1 for each condition. The participants will be stratified by aged into the age groups 12-14 years and 15-17 years respectively to secure an even age distribution across conditions. Additionally upon completing session 8 in the program, participants will be randomized to receive or not receive a booster session 12 weeks after finishing the intervention with an allocation ratio of 1:1. The design of the randomized trial is thus factorial including two factors: type of therapist feedback (factor 1) and booster or no booster (factor 2). Data will be collected with parent and adolescent questionnaires at five time points: pre-treatment, post-treatment and at follow-ups after 3, 6 and 12 months.
Masking Description: As the study concerns itself with psychotherapy and examines the difference in therapist support, it is practically impossible to blind participants and clinicians, and thus they are not blinded. The research team is involved in the day-to-day operation of the project, including the screening for suicidality, why blinding of the research team is also practically impossible with the current setup. However the analyzes of the trial results will be pseudo-anonymized, so that only the ID number appears on the data sheet in order to get as close to blinding as possible in relation to the research design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- iCBT with planned feedback (Experimental): Participants in this iCBT condition will receive written feedback from their therapist on assignments weekly. The participants will also be able to contact their assigned therapist through messages within the program and receive asynchronous support if needed. Participant depression and suicidality will also be continuously monitored using weekly questionnaires.
  Interventions: Behavioral: CoolMinds: Internet-based cognitive behavioral therapy (iCBT)
- iCBT with on-demand feedback (Experimental): Participants in the on-demand iCBT condition will not receive any planned contact with the therapist. However, the participants will be able to contact the therapist through messages within the program and receive asynchronous support if needed. The therapist will also be monitoring the participants' answers on questionnaires and assignments to ensure progress. Participant depression and suicidality will also be continuously monitored using weekly questionnaires.
  Interventions: Behavioral: CoolMinds: Internet-based cognitive behavioral therapy (iCBT)
- waitlist control (No Intervention): A waitlist control is included to compare the treatment conditions to a no-treatment condition and serves as a control for the effects of time and assessment on efficacy. Participants in the waitlist condition will be instructed to wait 14 weeks. After the 14-week period, participants will be offered iCBT treatment with planned therapist feedback and with elective modules. If participants do not wish to receive the iCBT treatment, they will receive help in finding another relevant treatment if needed.

INTERVENTIONS:
Behavioral: CoolMinds: Internet-based cognitive behavioral therapy (iCBT) — The intervention consists of 14 weeks of iCBT, where the main treatment components are psychoeducation, cognitive restructuring, exposure therapy, and relapse prevention. The program comprises eleven sessions for adolescents and ten sessions for parents to be completed simultaneously. The participants will have the opportunity to get therapist feedback during the treatment period, the therapist may spend a maximum of 15 minutes giving feedback per week per participant.
  Arms: iCBT with on-demand feedback; iCBT with planned feedback

SUMMARY:
The goal of the randomized controlled trial is to find out if the internet-based therapy (iCBT) intervention CoolMinds, is effective in helping adolescents with anxiety. The adolescents in the study are aged between 12 and 17 years of age, who live in the region of Southern Denmark. They must have an anxiety diagnosis according to the

Diagnostic and Statistical Manual-5 (DSM-5) criteria. The main questions it aims to answer are:

1. If getting anxiety treatment with CoolMinds will lead to a greater reduction in anxiety symptoms, compared to a waitlist.
2. What effect different degrees of therapist support have on the treatment.

Participants will be getting 14 weeks of the iCBT intervention CoolMinds, and they will be asked to answer questionnaires about their mental health before and after the treatment.

Researchers will compare three different groups, with 56 adolescents in each group. The first group will receive iCBT with weekly scheduled feedback. The second group will get iCBT with feedback whenever the adolescents ask for it. The last group will be on a waiting list for 14 weeks, before receiving treatment.

DETAILED DESCRIPTION:
Introduction

Among children and adolescents the most prevalent mental health conditions are anxiety disorders, with around 5-12% of youth in western countries fulfilling the criteria for an anxiety diagnosis. Evidence points to an increase in the prevalence of anxiety disorders during the transition from childhood to adolescence and from adolescence to adulthood up to age 30. Untreated anxiety disorders tend to chronify or become recurrent in the developmental course and persist into adulthood.

Cognitive behavioral therapy (CBT), in both individual and group format, is effective in treating young people with anxiety. Despite the existence of effective treatment options and the possible long-term consequences associated with untreated anxiety disorders in youth, it is estimated that less than 25% of children and adolescents with anxiety disorders receive professional help, with fewer receiving evidence-based treatment. Frequently mentioned barriers for adolescents opting to seek treatment include social stigma, shyness and fear of peer rejection, preference for self-reliance, confidentiality, privacy and anonymity concerns, worries concerning treatment costs, transportation or waiting times and limited availability of psychological treatment. Thus, it is of the utmost importance to consider these barriers when developing interventions to overcome these and thus increase treatment accessibility.

Internet-based cognitive behavioral therapy (iCBT) may be an effective alternative to face-to-face treatment, that can address some of the aforementioned barriers to treatment by providing greater flexibility, greater autonomy, reduced expenses, and eliminate travel time. To date, fourteen randomized controlled trials (RCTs) have evaluated iCBT programs in both children and adolescents with anxiety disorders. Four of these included predominantly or only adolescents and showed promising results with between group effect sizes ranging from d = 0.65-1.04 at follow-up.

Objectives

The primary aim of the present study is to examine the efficacy of an internet-delivered cognitive behavioral therapy intervention, CoolMinds, in adolescents aged 12-17 years, when delivered with planned feedback or on-demand feedback from a therapist compared to a waitlist control. Additionally, the study will explore the efficacy of delivering one booster session compared to none. It is hypothesized that:

1. CoolMinds will lead to a greater reduction in anxiety symptoms compared to the waitlist control.
2. The effect of CoolMinds will be independent of the degree of therapist support.

Design:

The study is designed as a superiority randomized controlled trial with the three conditions 1) iCBT with planned feedback 2) iCBT with on-demand feedback and 3) waitlist control. The allocation ratio is 1:1:1 for each condition. The participants will be stratified by aged into the age groups 12-14 years and 15-17 years respectively to secure an even age distribution across conditions. Additionally all participants that are active in the program for the first 8 weeks, will be randomized to receive or not receive a booster session 10 weeks after finishing the intervention with an allocation ratio of 1:1.

The study will be conducted at Center for Digital Psychiatry, an online clinic and research facility that is part of the psychiatric hospital in the region of southern Denmark, and at Center for Psychological Treatment of Children and Adolescents, a research and teaching center at Aarhus university, Denmark. All data will be collected from these two centers in Denmark.

Participants and recruitment:

All participants will have to register through a website to participate in the project. As part of the registration, the participants will have to fill out an initial screening questionnaire that assesses exclusion criteria. If an exclusion criteria is met, the participant will automatically be informed within the questionnaire that they are unable to participate and is given the choice to continue or discontinue their answering.

Data will be collected with a parent and adolescent questionnaire at five points: pre-treatment (T1), post-treatment (T2) and at follow-ups after 3, 6 and 12 months (T3, T4, T5). Participants in the waitlist control group will be offered guided iCBT with planned feedback at post-treatment (T2).

ELIGIBILITY:
Inclusion Criteria:

* Between 12 and 17 years of age.
* Have a principal anxiety diagnosis according to DSM-5 criteria.
* The ability to read and write Danish.
* Internet access.
* A parent able to participate in treatment alongside the adolescent.

Exclusion Criteria:

* Autism spectrum disorder.
* Attention deficit hyperactivity disorder.
* Psychotic symptoms.
* Bipolar disorder.
* Current suicidal ideation or self-mutilating behavior.
* Current alcohol or substance abuse.
* A score of 5 or above on ADIS
* Current eating disorder.
* Received CBT for an anxiety disorder within the past 12 months.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 168 (Estimated)
Dates: Start 2023-10-10 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
The Youth Online Diagnostic Assessment - Child and Parent Versions | Pre-treatment, immediately after treatment and at 3-month follow-up
  An online diagnostic assessment tool that assesses DSM-5 anxiety disorders and specific phobias based on the Anxiety and Related Disorders Interview Schedule for DSM-5, which is considered the golden standard.
Spence Children's Anxiety Scale- Child and Parent Versions | Pre-treatment, immediately after treatment and at 3- 6- 12-month follow-up
  A 44-item self-report questionnaire assessing anxiety symptoms of six different anxiety disorders in DSM-IV. The responses are scored on a 4 point scale ranging from 0 to 3, with a minimum score of 0 and a maximum score of 114, higher scores mean a higher level of anxiety.

SECONDARY OUTCOMES:
Child Anxiety Life Interference Scale- Child and Parent Version | Pre-treatment, immediately after treatment and at 3- 6- 12-month follow-up
  A 10-item self-report questionnaire assessing the impact of youth anxiety on various areas of life functioning such as school, extracurricular activities, family life and friendships. The responses are scored on a likert scale ranging from 0 to 4, with higher scores indicating higher anxiety life interference, minimum score is 0, maximum score is 36.
The Mood and Feelings Questionnaire- Child and Parent Version | Pre-treatment, immediately after treatment and at 3- 6- 12-month follow-up
  A 33-item self-report questionnaire assessing depression in youth, The responses are scored from 0 to 2, with higher scores suggest more severe depressive symptoms. Minimum score is 0, maximum score is 66.
Working Alliance Inventory - Short Form | Immediately after treatment and every 14 days during the treatment period
  A 12-item self-report questionnaire assessing the therapeutic alliance, the responses are scored from 1 to 7, minimum total score 12 to maximum total score of 84, higher scores reflect a more positive rating of working alliance.
Working Alliance Inventory for Online Interventions | Immediately after treatment
  A 36- items self-report questionnaire assessing the technical alliance, the responses are scored from 1 to 7, minimum total score 36 to maximum total score of 252, higher scores reflect a more positive rating of working alliance.

OTHER OUTCOMES:
Children´s Anxiety Scale | weekly questionnaire
  A 8-item abbreviated version of the Spence Children's Anxiety Scale containing 8 of the original 44-items. The responses are scored from 0 to 3, with a minimum total score of 0, to a maximum total score of 24. Higher scores mean a higher level of anxiety.
The Short Mood and Feelings questionnaire | Weekly questionnaire
  A 13-items self-report questionnaire with an added item about suicidal thoughts and ideation will assess the level of depressive symptoms and risk of suicide. The responses are scored from 0 to 2, with a minimum total score of 0, to a maximum total score of 26. with higher scores suggest more severe depressive symptoms.
EuroQol-5 Dimension Youth | Pre-treatment, immediately after treatment and at 3- 6- 12-month follow-up
  A 5-item self-report questionnaire assessing quality of life and self-rated health. The items cover five domains: mobility, selfcare, usual activities, pain/discomfort, and anxiety and depression. The responses are scored from 1 to 5, with a minimum total score of 5, to a maximum total score of 25. Higher score suggest problems with the different dimensions.
Client Satisfaction Questionnaire-8 | Immediately after treatment
  An 8-item questionnaire used to measure general satisfaction with a received treatment.The responses are scored from 1 to 4, with a minimum total score of 8, to a maximum total score of 32, with higher scores indicating greater satisfaction.
Systems Usability Scale | Immediately after treatment
  A 10-item questionnaire used to assess the subjective experience of usability of a higher score computer system. The responses are scored from 1 to 5, the participant´s scores for each question are converted to a new number, added together and then multiplied by 2.5 to make a scale with a minimum total score of 0, to a maximum total score of 100. A higher score indicates greater system usability.
Negative Effects Questionnaire | Immediately after treatment
  A 20-item questionnaire used to monitor the occurrence of negative effects in psychological treatments. The responses are scored from 0-4, with a minimum total score of 0, to a maximum total score of 80. A higher score indicates, more negative effects.
Sociodemographic measures | pre-treatment
  s will be gathered on parents regarding age, level of education, civil status, gender and primary caregiver in case of single parents. For the adolescents, information will be gathered regarding age and gender
Engagement | Immediately after treatment
  with the treatment will be measured objectively using the number of logins to the treatment program as well as number of words per message sent to the therapist and number of words per text box in the modules. This will be registered for both adolescents and parents.
Cost-effectiveness | Immediately after treatment
  Will be measured by self-report questionnaire about the number of days absent from school, if they have been in contact with self-paid psychiatrist or psychologist during the study and the use of communal services.
Cost-effectiveness | Immediately after treatment
  Will be measured by the time the parent and adolescent spent in the program, as well the therapists time spent on each patient.
The Anxiety Disorders Interview Schedule for Children | pre-treatment
  Depression will be measured oral during the clinical interview, with The Anxiety Disorders Interview Schedule for Children as The Youth Online Diagnostic Assessment depression module is not translated to Danish.

CONTACTS AND LOCATIONS:
Overall Officials: Kim Mathiasen, P.hd, Principal Investigator — Region of Southern Denmark
Locations (1):
- Centre for Digital Psychiatry, Odense, Region Syddanmark, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Data will be available for researches at Aarhus University, center for psychological treatment of children and adolescents. They will have access to study protocol, statistical analysis plan, informed consent form, clinical study report and analytical code.
  Data will also be stored on a server located in the Region of Southern Denmark. When the study is finished the data will be transferred to The Danish National Archives. Data are available upon reasonable request. Restrictions apply to the availability of data and approval is needed from Danish Data Protection Agency and or The Danish National Archives.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data is available for researchers from Aarhus University, center for psychological treatment of children and adolescents during and after the study is finished.
  For other the data will become available after the study is finished
Access Criteria: There have been made an data sharing agreement between Aarhus University, center for psychological treatment of children and adolescents and the region of southern Denmark, the agreement must be followed
  Restrictions apply to the availability of data and approval is needed from Danish Data Protection Agency and or The Danish National Archives.

REFERENCES:
- [Background] Angold, A., Costello, E. J., Messer, S. C., & Pickles, A. (1995). Development of a short questionnaire for use in epidemiological studies of depression in children and adolescents. International Journal of Methods in Psychiatric Research.
- [Background] Arendt K, Hougaard E, Thastum M. Psychometric properties of the child and parent versions of Spence children's anxiety scale in a Danish community and clinical sample. J Anxiety Disord. 2014 Dec;28(8):947-56. doi: 10.1016/j.janxdis.2014.09.021. Epub 2014 Oct 16. PMID 25445085
- [Background] Attkisson, C. C., & Greenfield, T. K. (1994). Client Satisfaction Questionnaire-8 and Service Satisfaction Scale-30.
- [Background] Beesdo K, Knappe S, Pine DS. Anxiety and anxiety disorders in children and adolescents: developmental issues and implications for DSM-V. Psychiatr Clin North Am. 2009 Sep;32(3):483-524. doi: 10.1016/j.psc.2009.06.002. PMID 19716988
- [Background] Berg M, Rozental A, de Brun Mangs J, Nasman M, Stromberg K, Viberg L, Wallner E, Ahman H, Silfvernagel K, Zetterqvist M, Topooco N, Capusan A, Andersson G. The Role of Learning Support and Chat-Sessions in Guided Internet-Based Cognitive Behavioral Therapy for Adolescents With Anxiety: A Factorial Design Study. Front Psychiatry. 2020 Jun 10;11:503. doi: 10.3389/fpsyt.2020.00503. eCollection 2020. PMID 32587533
- [Background] Brooke, J. (1996). SUS: A "quick and dirty" usability scale. In J. B. W. Thomas, B. (Ed.), Usability evaluation in industry (pp. 189-194). London, UK: Taylor & Francis.
- [Background] Costello EJ, Egger HL, Angold A. The developmental epidemiology of anxiety disorders: phenomenology, prevalence, and comorbidity. Child Adolesc Psychiatr Clin N Am. 2005 Oct;14(4):631-48, vii. doi: 10.1016/j.chc.2005.06.003. PMID 16171696
- [Background] Daviss WB, Birmaher B, Melhem NA, Axelson DA, Michaels SM, Brent DA. Criterion validity of the Mood and Feelings Questionnaire for depressive episodes in clinic and non-clinic subjects. J Child Psychol Psychiatry. 2006 Sep;47(9):927-34. doi: 10.1111/j.1469-7610.2006.01646.x. PMID 16930387
- [Background] Eg J, Bilenberg N, Costello EJ, Wesselhoeft R. Self- and parent-reported depressive symptoms rated by the mood and feelings questionnaire. Psychiatry Res. 2018 Oct;268:419-425. doi: 10.1016/j.psychres.2018.07.016. Epub 2018 Jul 22. PMID 30130708
- [Background] Gulliver A, Griffiths KM, Christensen H. Perceived barriers and facilitators to mental health help-seeking in young people: a systematic review. BMC Psychiatry. 2010 Dec 30;10:113. doi: 10.1186/1471-244X-10-113. PMID 21192795
- [Background] Herrero R, Vara MD, Miragall M, Botella C, Garcia-Palacios A, Riper H, Kleiboer A, Banos RM. Working Alliance Inventory for Online Interventions-Short Form (WAI-TECH-SF): The Role of the Therapeutic Alliance between Patient and Online Program in Therapeutic Outcomes. Int J Environ Res Public Health. 2020 Aug 25;17(17):6169. doi: 10.3390/ijerph17176169. PMID 32854381
- [Background] Hvidt, J. C. S., Christensen, L. F., Sibbersen, C., Helweg-Jørgensen, S., Hansen, J. P., & Lichtenstein, M. B. (2020). Translation and Validation of the System Usability Scale in a Danish Mental Health Setting Using Digital Technologies in Treatment Interventions. International journal of human-computer interaction, 36(8), 709-716. doi:10.1080/10447318.2019.1680922
- [Background] James AC, Reardon T, Soler A, James G, Creswell C. Cognitive behavioural therapy for anxiety disorders in children and adolescents. Cochrane Database Syst Rev. 2020 Nov 16;11(11):CD013162. doi: 10.1002/14651858.CD013162.pub2. PMID 33196111
- [Background] Jolstedt M, Wahlund T, Lenhard F, Ljotsson B, Mataix-Cols D, Nord M, Ost LG, Hogstrom J, Serlachius E, Vigerland S. Efficacy and cost-effectiveness of therapist-guided internet cognitive behavioural therapy for paediatric anxiety disorders: a single-centre, single-blind, randomised controlled trial. Lancet Child Adolesc Health. 2018 Nov;2(11):792-801. doi: 10.1016/S2352-4642(18)30275-X. Epub 2018 Sep 18. PMID 30241993
- [Background] Keller MB, Lavori PW, Wunder J, Beardslee WR, Schwartz CE, Roth J. Chronic course of anxiety disorders in children and adolescents. J Am Acad Child Adolesc Psychiatry. 1992 Jul;31(4):595-9. doi: 10.1097/00004583-199207000-00003. PMID 1644719
- [Background] Kessler RC, Berglund P, Demler O, Jin R, Merikangas KR, Walters EE. Lifetime prevalence and age-of-onset distributions of DSM-IV disorders in the National Comorbidity Survey Replication. Arch Gen Psychiatry. 2005 Jun;62(6):593-602. doi: 10.1001/archpsyc.62.6.593. PMID 15939837
- [Background] Khanna MS, Kendall PC. Computer-assisted cognitive behavioral therapy for child anxiety: results of a randomized clinical trial. J Consult Clin Psychol. 2010 Oct;78(5):737-45. doi: 10.1037/a0019739. PMID 20873909
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Leigh E, Clark DM. Internet-delivered therapist-assisted cognitive therapy for adolescent social anxiety disorder (OSCA): a randomised controlled trial addressing preliminary efficacy and mechanisms of action. J Child Psychol Psychiatry. 2023 Jan;64(1):145-155. doi: 10.1111/jcpp.13680. Epub 2022 Aug 9. PMID 35943064
- [Background] March S, Spence SH, Donovan CL. The efficacy of an internet-based cognitive-behavioral therapy intervention for child anxiety disorders. J Pediatr Psychol. 2009 Jun;34(5):474-87. doi: 10.1093/jpepsy/jsn099. Epub 2008 Sep 15. PMID 18794187
- [Background] McLellan LF, Kangas M, Rapee RM, Iverach L, Wuthrich VM, Hudson JL, Lyneham HJ. The Youth Online Diagnostic Assessment (YODA): Validity of a New Tool to Assess Anxiety Disorders in Youth. Child Psychiatry Hum Dev. 2021 Apr;52(2):270-280. doi: 10.1007/s10578-020-01007-3. PMID 32440754
- [Background] Merikangas KR, He JP, Burstein M, Swanson SA, Avenevoli S, Cui L, Benjet C, Georgiades K, Swendsen J. Lifetime prevalence of mental disorders in U.S. adolescents: results from the National Comorbidity Survey Replication--Adolescent Supplement (NCS-A). J Am Acad Child Adolesc Psychiatry. 2010 Oct;49(10):980-9. doi: 10.1016/j.jaac.2010.05.017. Epub 2010 Jul 31. PMID 20855043
- [Background] Merikangas KR, He JP, Burstein M, Swendsen J, Avenevoli S, Case B, Georgiades K, Heaton L, Swanson S, Olfson M. Service utilization for lifetime mental disorders in U.S. adolescents: results of the National Comorbidity Survey-Adolescent Supplement (NCS-A). J Am Acad Child Adolesc Psychiatry. 2011 Jan;50(1):32-45. doi: 10.1016/j.jaac.2010.10.006. Epub 2010 Dec 3. PMID 21156268
- [Background] Messer, S. C., Angold, A., Costello, E. J., Loeber, R., Van Kammen, W., & Stouthamer-Loeber, M. (1995). Development of a short questionnaire for use in epidemiological studies of depression in children and adolescents: Factor composition and structure across development. International Journal of Methods in Psychiatric Research, 5, 251-262.
- [Background] Musiat P, Goldstone P, Tarrier N. Understanding the acceptability of e-mental health--attitudes and expectations towards computerised self-help treatments for mental health problems. BMC Psychiatry. 2014 Apr 11;14:109. doi: 10.1186/1471-244X-14-109. PMID 24725765
- [Background] Nearchou FA, Bird N, Costello A, Duggan S, Gilroy J, Long R, McHugh L, Hennessy E. Personal and perceived public mental-health stigma as predictors of help-seeking intentions in adolescents. J Adolesc. 2018 Jul;66:83-90. doi: 10.1016/j.adolescence.2018.05.003. Epub 2018 May 23. PMID 29800758
- [Background] Nordh M, Wahlund T, Jolstedt M, Sahlin H, Bjureberg J, Ahlen J, Lalouni M, Salomonsson S, Vigerland S, Lavner M, Ost LG, Lenhard F, Hesser H, Mataix-Cols D, Hogstrom J, Serlachius E. Therapist-Guided Internet-Delivered Cognitive Behavioral Therapy vs Internet-Delivered Supportive Therapy for Children and Adolescents With Social Anxiety Disorder: A Randomized Clinical Trial. JAMA Psychiatry. 2021 Jul 1;78(7):705-713. doi: 10.1001/jamapsychiatry.2021.0469. PMID 33978699
- [Background] Polanczyk GV, Salum GA, Sugaya LS, Caye A, Rohde LA. Annual research review: A meta-analysis of the worldwide prevalence of mental disorders in children and adolescents. J Child Psychol Psychiatry. 2015 Mar;56(3):345-65. doi: 10.1111/jcpp.12381. Epub 2015 Feb 3. PMID 25649325
- [Background] Reardon T, Harvey K, Creswell C. Seeking and accessing professional support for child anxiety in a community sample. Eur Child Adolesc Psychiatry. 2020 May;29(5):649-664. doi: 10.1007/s00787-019-01388-4. Epub 2019 Aug 13. PMID 31410579
- [Background] Rickwood DJ, Braithwaite VA. Social-psychological factors affecting help-seeking for emotional problems. Soc Sci Med. 1994 Aug;39(4):563-72. doi: 10.1016/0277-9536(94)90099-x. PMID 7973856
- [Background] Rickwood DJ, Deane FP, Wilson CJ. When and how do young people seek professional help for mental health problems? Med J Aust. 2007 Oct 1;187(S7):S35-9. doi: 10.5694/j.1326-5377.2007.tb01334.x. PMID 17908023
- [Background] Spence SH, Donovan CL, March S, Gamble A, Anderson RE, Prosser S, Kenardy J. A randomized controlled trial of online versus clinic-based CBT for adolescent anxiety. J Consult Clin Psychol. 2011 Oct;79(5):629-42. doi: 10.1037/a0024512. PMID 21744945
- [Background] Spence SH, Donovan CL, March S, Kenardy JA, Hearn CS. Generic versus disorder specific cognitive behavior therapy for social anxiety disorder in youth: A randomized controlled trial using internet delivery. Behav Res Ther. 2017 Mar;90:41-57. doi: 10.1016/j.brat.2016.12.003. Epub 2016 Dec 8. PMID 27988427
- [Background] Spence SH, Holmes JM, March S, Lipp OV. The feasibility and outcome of clinic plus internet delivery of cognitive-behavior therapy for childhood anxiety. J Consult Clin Psychol. 2006 Jun;74(3):614-21. doi: 10.1037/0022-006X.74.3.614. PMID 16822117
- [Background] Stallard P, Velleman S, Richardson T. Computer Use and Attitudes Towards Computerised Therapy Amongst Young People and Parents Attending Child and Adolescent Mental Health Services. Child Adolesc Ment Health. 2010 May;15(2):80-84. doi: 10.1111/j.1475-3588.2009.00540.x. Epub 2009 Sep 24. PMID 32847246
- [Background] Stjerneklar S, Hougaard E, McLellan LF, Thastum M. A randomized controlled trial examining the efficacy of an internet-based cognitive behavioral therapy program for adolescents with anxiety disorders. PLoS One. 2019 Sep 18;14(9):e0222485. doi: 10.1371/journal.pone.0222485. eCollection 2019. PMID 31532802
- [Background] Storch EA, Salloum A, King MA, Crawford EA, Andel R, McBride NM, Lewin AB. A RANDOMIZED CONTROLLED TRIAL IN COMMUNITY MENTAL HEALTH CENTERS OF COMPUTER-ASSISTED COGNITIVE BEHAVIORAL THERAPY VERSUS TREATMENT AS USUAL FOR CHILDREN WITH ANXIETY. Depress Anxiety. 2015 Nov;32(11):843-52. doi: 10.1002/da.22399. Epub 2015 Sep 14. PMID 26366886
- [Background] Vigerland S, Ljotsson B, Thulin U, Ost LG, Andersson G, Serlachius E. Internet-delivered cognitive behavioural therapy for children with anxiety disorders: A randomised controlled trial. Behav Res Ther. 2016 Jan;76:47-56. doi: 10.1016/j.brat.2015.11.006. Epub 2015 Nov 19. PMID 26649465
- [Background] Waite P, Marshall T, Creswell C. A randomized controlled trial of internet-delivered cognitive behaviour therapy for adolescent anxiety disorders in a routine clinical care setting with and without parent sessions. Child Adolesc Ment Health. 2019 Sep;24(3):242-250. doi: 10.1111/camh.12311. Epub 2019 Mar 6. PMID 32677216
- [Background] Wang PS, Angermeyer M, Borges G, Bruffaerts R, Tat Chiu W, DE Girolamo G, Fayyad J, Gureje O, Haro JM, Huang Y, Kessler RC, Kovess V, Levinson D, Nakane Y, Oakley Brown MA, Ormel JH, Posada-Villa J, Aguilar-Gaxiola S, Alonso J, Lee S, Heeringa S, Pennell BE, Chatterji S, Ustun TB. Delay and failure in treatment seeking after first onset of mental disorders in the World Health Organization's World Mental Health Survey Initiative. World Psychiatry. 2007 Oct;6(3):177-85. PMID 18188443
- [Background] Wuthrich VM, Rapee RM, Cunningham MJ, Lyneham HJ, Hudson JL, Schniering CA. A randomized controlled trial of the Cool Teens CD-ROM computerized program for adolescent anxiety. J Am Acad Child Adolesc Psychiatry. 2012 Mar;51(3):261-70. doi: 10.1016/j.jaac.2011.12.002. Epub 2012 Jan 21. PMID 22365462
- [Background] Zhou X, Zhang Y, Furukawa TA, Cuijpers P, Pu J, Weisz JR, Yang L, Hetrick SE, Del Giovane C, Cohen D, James AC, Yuan S, Whittington C, Jiang X, Teng T, Cipriani A, Xie P. Different Types and Acceptability of Psychotherapies for Acute Anxiety Disorders in Children and Adolescents: A Network Meta-analysis. JAMA Psychiatry. 2019 Jan 1;76(1):41-50. doi: 10.1001/jamapsychiatry.2018.3070. PMID 30383099
- [Derived] Skaarnes H, Sorensen NM, Wisnewski AH, Lomholt JJ, Thastum M, McLellan L, Mathiasen K. Internet-based cognitive behavioral intervention for adolescents with anxiety disorders: a study protocol for a parallel three armed randomized controlled trial. Trials. 2024 Oct 13;25(1):674. doi: 10.1186/s13063-024-08511-0. PMID 39396991